CLINICAL TRIAL: NCT02751996
Title: A Phase 2, Open-label, Randomized, Two-part, Multiple Dose Study Evaluating the Safety, Pharmacokinetics, and Antiviral Efficacy of SB 9200 in Subjects Infected With Chronic Hepatitis B Virus
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Antiviral Efficacy of SB 9200 in Subjects Infected With Chronic HBV
Acronym: ACHIEVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: F-star Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBP-9200-HBV-201
Record Dates: First submitted 2016-04-06; First posted 2016-04-26 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis B; Hepatitis, Viral
Keywords: Chronic Hepatitis; HBV; Double blind
MeSH Terms: conditions — Hepatitis B; Hepatitis; Hepatitis, Chronic | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Part A Cohort 1: 25mg SB 9200 (Active Comparator): Part A Cohort 1: 25mg SB 9200. After 12 weeks of SB 9200 this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: SB 9200
- Part A Cohort 1: 25mg Placebo (Placebo Comparator): Part A Cohort 1: 25mg Placebo. After 12 weeks of Placebo this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: Placebo
- Part A Cohort 2: 50mg SB 9200 (Active Comparator): Part A Cohort 2: 50mg SB 9200. After 12 weeks of SB 9200 this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: SB 9200
- Part A Cohort 2: 50mg Placebo (Placebo Comparator): Part A Cohort 2: 50mg Placebo. After 12 weeks of Placebo this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: Placebo
- Part A Cohort 3: 100mg SB 9200 (Active Comparator): Part A Cohort 3: 100mg SB 9200. After 12 weeks of SB 9200 this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: SB 9200
- Part A Cohort 3: 100mg Placebo (Placebo Comparator): Part A Cohort 3: 100mg Placebo. After 12 weeks of Placebo this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: Placebo
- Part A Cohort 4: 200mg SB 9200 (Active Comparator): Part A Cohort 4: 200mg SB 9200. After 12 weeks of SB 9200 this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: SB 9200
- Part A Cohort 4: 200mg Placebo (Placebo Comparator): Part A Cohort 4: 200mg Placebo. After 12 weeks of Placebo this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: Placebo
- Part B: SB 9200 with tenofovir (Active Comparator): Part B: SB 9200 selected dose from Part A administered in combination with tenofovir 300 mg qd. After 12 weeks of SB 9200 this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: SB 9200
- Part B: Tenofovir 300 mg (Active Comparator): Part B: Tenofovir 300 mg qd monotherapy. After 12 weeks of SB 9200 this medication will be stopped. From weeks 12 - 24 patients will be given 12 weeks of Tenofovir (current standard of care)
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: SB 9200 — SB 9200
  Other Names: SB9200
  Arms: Part A Cohort 1: 25mg SB 9200; Part A Cohort 2: 50mg SB 9200; Part A Cohort 3: 100mg SB 9200; Part A Cohort 4: 200mg SB 9200; Part B: SB 9200 with tenofovir
Drug: Placebo
  Arms: Part A Cohort 1: 25mg Placebo; Part A Cohort 2: 50mg Placebo; Part A Cohort 3: 100mg Placebo; Part A Cohort 4: 200mg Placebo
Drug: Tenofovir
  Arms: Part B: Tenofovir 300 mg

SUMMARY:
This is a Phase 2, open-label,randomized, multiple dose, varied administration regimen study with 2 parts (Parts A and B) in Subjects Infected with Chronic Hepatitis B Virus

DETAILED DESCRIPTION:
This is a Phase 2, open-label, randomized, multiple dose, varied administration regimen study with 2 parts (Parts A and B).

Part A will utilize an ascending dose cohort design with sequential cohorts. Each cohort will be evaluated by the DSMB for safety. Additional cohorts may be added by the DSMB to determine doses of SB 9200 that exhibit significant antiviral response and safety.

Approximately 80 subjects will be assigned sequentially to 1 of the following dosing cohorts (20 subjects per cohort) and randomized in a 4:1 ratio (active:placebo) within each cohort. Randomization will be stratified so that no more than 2 HBeAg positive subjects will be assigned to receive placebo.

* SB 9200 25 mg or matching placebo administered qd
* SB 9200 50 mg or matching placebo administered qd
* SB 9200 100 mg or matching placebo administered qd
* SB 9200 200 mg or matching placebo administered qd

After informed consent is obtained, subjects will enter a Screening period, which will last up to 28 days. Once all eligibility criteria are confirmed and the subject is randomized, subjects will receive the IP or placebo as a 2-week supply of capsules/tablets. All randomized subjects will receive the IP or matching placebo for a total of 12 weeks. All subjects will then receive tenofovir 300 mg qd for an additional 12 weeks of treatment.

Subjects will start the treatment period on Day 1. The PK samples will be collected on Day 1 at predose, 30 minutes, 1, 2, 4, 6, and 24 hours (predose the following day). At Week 6, the same sampling times will be used to collect PK samples from the subjects to collect steady state PK data. Subjects will return biweekly for the entire 12-week IP treatment period, except when beginning IP administration when subjects will be seen weekly, for safety assessments including physical examination and laboratory sample analysis of chemistry, hematology, and urine. Sample collection for efficacy (HBV DNA, HBsAg, HBeAg, hepatitis B envelope antibody [HBeAb], HBV RNA, and HBV resistance) will be collected as indicated in the Schedule of Events. A sample for genotyping will be collected at Day 1. Samples for Locarnini biomarkers and other biomarkers will also occur at Day 1; Weeks 2, 4, 8, 12, and 14; and at the End of Study Visit. Samples for cytokine levels will be collected at Day 1, Week 6, and Week 12. At Week 12, the end of IP administration, all subjects will return to the clinic and be administered IP and 300 mg tenofovir. Samples will be collected to explore the potential of a drug-drug interaction between SB 9200 and tenofovir. All subjects will have a predose PK sample then take the last dose of IP/placebo together with their first dose of tenofovir. The PK samples will then be collected for SB 9200 and tenofovir at 30 minutes,and 1, 2, 4, 6, and 24 hours. Thereafter, the subjects will receive only tenofovir 300 mg qd for an additional 12 weeks as 4-week supplies. All subjects will return to the clinic at Weeks 13, 14, 16, 20, and 24. Subjects will have safety assessments including symptom-directed physical examinations and safety hematology, biochemistry, and virological studies performed at these visits.

At Week 24, all subjects will have completed the study Part A (or Part B, as applicable).

Part B will be an open-label, randomized, combination therapy design consisting of multiple cohorts. The study is designed to evaluate the safety, tolerability, and antiviral response in subjects treated for 12 weeks with a dose of SB 9200 selected from Part A that exhibits significant antiviral response and safety when administered in combination with tenofovir 300 mg qd (Cohort 1) or with tenofovir 300 mg qd monotherapy alone (Cohort 2). All subjects will then continue in the study for an additional 12 weeks with tenofovir alone. Randomization between the 2 initial cohorts will be conducted using a 3:1 ratio resulting in 30 subjects being allocated to SB 9200 in combination with tenofovir (Cohort 1) and 10 subjects being allocated to tenofovir monotherapy (Cohort 2). No cohort can enroll more than 60% of either hepatitis e antigen negative or hepatitis e antigen positive subjects.

Part B will utilize an adaptive design. The first 2 cohorts of Part B may start concurrently to Part A at any time after a dose has been selected from Part A. SB 9200 doses for which all subjects have not completed the initial 12 weeks monotherapy of SB 9200 from Part A and demonstrated safety of IP will not be selected to be administered in combination with tenofovir during Part B.

The first 2 cohorts will randomize concurrently using a 3:1 ratio.

* Cohort 1: 30 subjects will receive SB 9200 selected dose #1 from Part A administered in combination with tenofovir 300 mg qd.
* Cohort 2: 10 subjects will receive tenofovir 300 mg qd monotherapy.

Based on the results of Part A completed and ongoing cohorts and Part B first cohort, up to 2 additional cohorts for which the dose of SB 9200 will be either escalated or de-escalated may be opened to enrollment:

* Cohort 3: 30 subjects will receive SB 9200 selected dose #2 from Part A administered in combination with tenofovir 300 mg qd.
* Cohort 4: 30 subjects will receive SB 9200 selected dose #3 from Part A administered in combination with tenofovir 300 mg qd.

Subjects will be enrolled into the Screening period, which will last up to 28 days. Once all eligibility criteria are confirmed, subjects will receive the IP as a 2-week supply of capsules/tablets and tenofovir as a 4-week supply. Subjects will be required to take the IP per protocol for 12 weeks. Subjects will return biweekly for the entire 12-week IP treatment period, except when beginning IP administration when subjects will be seen weekly, for safety assessments including physical examination and laboratory sample analysis of chemistry, hematology, and urine. Samples for Locarnini biomarkers will also occur at Day 1; Weeks 2, 4, 6, 12, and 14; and at the End of Study Visit. Sample collection for cytokine levels and other biomarkers of immune response and plasma samples will also occur at predose on Day 1 and at Weeks 6,12 and 24. The PK samples will be collected on Day 1 at predose, 30 minutes, and 1, 2, 4, 6, and 24 hours (predose the following day). At Week 12, the same sampling times will be used to collect PK samples from the subjects to collect steady state PK data. Sample collection for population PK analysis will also be collected before IP administration at Weeks 4 and 8. Urinary PK will be collected on Day 1 and Week 12 predose, 6 hours, and 24 hours (predose the following day).

At Week 12, all subjects will be administered tenofovir 300 mg qd for an additional 12 weeks as 4-week supplies. All subjects will return to the clinic at Weeks 13, 14, 16, 20, and 24. Subjects will have safety assessments including symptom-directed physical examinations and safety hematology, biochemistry, and virological studies performed at these visits.

Safety reporting for each subject in each cohort will continue after the subject first consents to participate in the study through the 24 week duration of the study or through the Extension Period until 30 days after the last dose is administered.

At Week 24, all subjects will have completed the study Part A (or Part B, as applicable).

Extension Period:

Any subject who completes Part A or Part B may be eligible to take part in a 12-month Extension Period. Before any study-related procedures are performed, the subjects will have all study procedures explained to them, including information regarding the nature of the study, and subjects must sign an informed consent/assent form. During the Extension Period, subjects will receive tenofovir and return for visits every 3 months with laboratory tests of liver function and virological efficacy including HBsAg, HBeAg, HBeAb, and HBV DNA. No further study-related testing will be performed. Subjects who undergo full termination from the study during Part A or Part B will not be eligible to enroll into the extension study.

Safety reporting for each subject in each cohort will continue after the subject first consents to participate in the study through the 24-week duration of the study or through the Extension Period until 30 days after the last dose is administered.

ELIGIBILITY:
Inclusion Criteria:

1. Documented evidence of chronic HBV infection (eg, HBsAg positive for at least 6 months or HBV DNA positive for at least 6 months). In the absence of documented evidence of HBsAg or HBV DNA, the subject must be HBsAg positive, and anti-HBc (IgM) negative at Screening.
2. Not on any antiviral medications for at least 6 months. If a subject is HBeAg negative, they will be eligible if they have not received antiviral medications for at least 3 months. Antiviral medications include lamivudine, telbivudine, adefovir, tenofovir, entecavir, IFN therapies of any type, and all other medications with potential antiviral activity.
3. HBV DNA > 2000 IU/mL for HBeAg-negative subjects and > 20000 IU/mL for HBeAg-positive subjects at Screening
4. ALT > ULN, but < 5 x the ULN and ≤ 200 U/L
5. Ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) within 3 months of randomization date with no evidence of hepatocellular carcinoma
6. Must be willing and able to comply with all study requirements
7. Negative urine or serum pregnancy test (for women of childbearing potential [WOCBP]) documented within the 24-hour period prior to the first dose of test drug. If the urine pregnancy test is positive, a follow-up serum test is required for confirmation. Additionally, all fertile males with partners of childbearing age and females must be using reliable contraception during the study and for 3 months after treatment completion. All fertile males must also refrain from sperm donation while on IP and for 3 months after completion of IP.
8. Must have the ability to understand and sign a written ICF; consent must be obtained prior to initiation of study procedures

Inclusion Criteria for Extension Period:

Subjects who meet all of the following inclusion criteria may be eligible to be enrolled into the Extension Period:

1. Signed informed consent form
2. Subject was randomized in Part A or Part B

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Any prior liver biopsy evidence of metavir F3 or F4 disease
2. Any history of decompensation of liver disease including history of ascites, encephalopathy, or varices
3. Evidence of cirrhosis as defined by Fibroscan at the Screening Visit of ≥ 8 kilopascals (kPa) or both a Fibrotest ≥ 0.65 and AST:platelet ratio index (APRI) ≥ 1.0 (subjects will not be excluded if only 1 of the Fibrotest or APRI result is higher than allowed) or have had evidence of Metavir F3-F4 on liver biopsy at any time.
4. Laboratory parameters not within defined thresholds: white blood cells (WBC) < 4000 cells/µL, (SI unit < 4.0 × 109/L), hemoglobin (HgB) < 12 g/dL (SI unit < 120 g/L) for females, < 13 g/dL (SI unit < 130 g/L) for males, platelets < 130,000 per µL, (SI unit < 130 × 109/L), albumin < 3.5 g/dL,(SI unit < 35 g/L), international normalized ratio (INR) > 1.5, total bilirubin > 1.2 mg/dL, (SI unit > 20.52 µmol/L), or alpha-fetoprotein (AFP) > 50 ng/mL (SI unit > 180.25 nmol/L). Subjects with an elevated indirect bilirubin and known Gilbert's disease can be included if direct bilirubin is within normal limits. Subjects with an AFP > 50 ng/mL but ˂ 500 ng/mL can be included if computed tomography (CT) scan or magnetic resonance imaging (MRI) performed within 3 months shows no evidence of hepatocellular carcinoma
5. Creatinine > 1.2 mg/dL, (SI unit > 106.08 µmol/L), creatinine clearance < 50 mL/min, (SI unit < 0.83 L/s/m2)
6. Co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis D virus
7. Evidence or history of hepatocellular carcinoma
8. Malignancy within 5 years prior to Screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible.
9. Significant cardiovascular, pulmonary, or neurological disease
10. Received solid organ or bone marrow transplant
11. Received within 3 months of Screening or expected to receive prolonged therapy with immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal antibody, IFN)
12. Subjects currently taking medication(s) that are transported through organic anion transporting polypeptide 1 (OATP1) including, but not limited to, atazanavir, rifampin, cyclosporine, eltrombopag, gemfibrozil, lopinavir/ritonavir, and saquinavir
13. Use of another investigational agent within 3 months of Screening
14. Current alcohol or substance abuse judged by the Investigator to potentially interfere with compliance
15. Females who are pregnant or may wish to become pregnant during the study
16. If the Investigator believes the prospective subject will not be able to comply with the requirements of the protocol and complete the study
17. Any medical condition, in the opinion of the Investigator, that could interfere with evaluation of the study objectives or safety of the subjects

Exclusion Criteria for Extension Period Subjects who meet any of the following exclusion criteria are not to be enrolled into the Extension Period:

1. Any condition, comorbidity, or laboratory abnormality that, based on the package insert of tenofovir or in the opinion of the Investigator, excludes the subject
2. Subjects who were withdrawn from Part A or Part B due to an AE or serious adverse event (SAE) related to the use of tenofovir
3. Participation in any other interventional study
4. Subject fully terminated from Part A or Part B

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Part A: Proportion of subjects reporting an adverse event (AE) and HBV DNA decline | 12 weeks
  The primary endpoint for safety and efficacy in Part A is the proportion of subjects reporting an adverse event (AE) or experiencing a clinically significant AE or laboratory abnormality from baseline (Randomisation) to end of SB 9200 treatment (12 weeks) and change from baseline to Week 12 in Log10 HBV DNA.
Part B: Proportion of subjects reporting an adverse event (AE) and hepatitis B surface antigen decline | 12 weeks
  The primary endpoints for safety and efficacy in Part B is the proportion of subjects reporting an adverse event (AE) or experiencing a clinically significant AE or laboratory abnormality from baseline (Randomisation) to end of SB 9200 treatment (12 weeks) and the proportion of subjects with hepatitis B surface antigen decline (12 weeks)

SECONDARY OUTCOMES:
Maximum observed plasma SB 9200 plasma concentration (Cmax) and determination of pharmacokineticPK parameters for SB 9200 and, Rp -SB 9000, and Sp SB 9000 (Parts A and B) | 0 - 24 hours
Change in serum HBV DNA, HBsAg, and HBV RNA at 2, 4, 8, 12, 14, and 24 weeks (Part A) | 2, 4, 8, 12, 14, and 24 weeks
Change in serum HBV DNA, HBsAg, and HBV RNA at 2, 4, 6, 12, 14, and 24 weeks (Part B) | 2, 4, 6, 12, 14, and 24 weeks
Change in HBeAg in log10 IU/mL from Baseline to Weeks 2, 4, 8, 12, 14, and 24 (Part A) | Weeks 2, 4, 8, 12, 14, and 24 weeks
Change in HBeAg in log10 IU/mL from Baseline to Weeks 2, 4, 6, 12, 14, and 24 (Part B) | 2, 4, 6, 12, 14, and 24 weeks
Proportion of subjects with HBeAg or HBsAg loss and seroconversion at Weeks 2, 4, 8, 12, 14, and 24 (Part A) | 2, 4, 8, 12, 14, and 24 weeks
Proportion of subjects with HBeAg or HBsAg loss and seroconversion at Weeks 2, 4, 6, 12, 14, and 24 (Part B) | 2, 4, 6, 12, 14, and 24 weeks
Proportion of subjects with HBsAg ≥ 1 log10 reduction from Baseline to Week 12 (Part B) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Macfarlane, Study Director — SBP Sr. Director of Clinical Operations
Locations (17):
- Canada (5):
  - Spring Bank Pharma Research site, Calgary, Alberta
  - Spring Bank Pharma Research site, Vancouver, British Columbia
  - Spring Bank Pharma Research Site, London, Ontario
  - Spring Bank Pharma Research site, Toronto, Ontario
  - Spring Bank Pharma Research site, Vaughan, Ontario
- Hong Kong (2):
  - Spring Bank Pharma Research site, Hong Kong
  - Spring Bank Pharma Research site, Shatin
- South Korea (6):
  - Spring Pharma Research Site, Chuncheon, Gangwon-do
  - Spring Bank Pharma Research site, Yangsan, Gyeongsangnam-do
  - Spring Bank Pharma Research site, Busan
  - Spring Bank Pharma Research Site, Daegu
  - Spring Bank Pharma Research site, Goyang-si
  - Spring Bank Pharma Research site, Seoul
- Taiwan (4):
  - Spring Bank Pharma Research Site, Chia-Yi City
  - Spring Bank Pharma Research Site, New Taipei City
  - Spring Bank Pharma Research Site, Taipei
  - Spring Bank Pharma Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: No
No plan to share data at this stage